CLINICAL TRIAL: NCT01342679
Title: A Study of Complete Molecular Response for Chronic Myeloid Leukemia in Chronic Phase Patients, Treated With Dasatinib
Acronym: CMR-CML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kanto CML Study Group (Other)
Collaborators: Epidemiological and Clinical Research Information Network (Other)
Responsible Party: Hisashi Sakamaki, Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCSG-02
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Myeloid Leukemia
Keywords: chronic myeloid leukemia; dasatinib; complete molecular response
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dasatinib (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — 100mg QD
  Other Names: BMS-354825

SUMMARY:
The purpose of this study is to evaluate complete molecular response of Dasatinib in patients for Philadelphia chromosome-positive chronic myeloid leukemia

ELIGIBILITY:
Inclusion Criteria:

* Chronic Myeloid Leukemia in the Chronic Phase
* 20 years old over
* ECOG performance status (PS) score 0-2
* Patients for major molecular response (MMR) with no CMR
* Adequate organ function (hepatic, renal and lung)
* Signed written informed consent

Exclusion Criteria:

* A case with the double cancer of the activity
* Women who are pregnant or breastfeeding
* The case of Pleural effusion clearly
* Patients with complications or a history of severe or uncontrolled cardiovascular failure following

  * have a Myocardial infarction within 6 months
  * have an Angina within 3 months
  * have a Congestive heart failure within 3 months
  * have a suspected congenital QT syndrome
  * have a QTc interval of more than 450msec at baseline
* A serious uncontrolled medical disorder that would impair the ability of the subjects to receive protocol therapy
* Prior treatment with dasatinib
* Subjects with T315I, F317L and V299L BCR-ABL point mutations

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Rate of complete molecular response (CMR) after treatment with dasatinib | at 12 months

SECONDARY OUTCOMES:
Dasatinib of dose intensity | at 12 months
Expansions rate of large granular lymphocyte | at 12 months
Progression free survival | at 12 months
Number of Participants with Adverse Events | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chikashi Yoshida, MD, PhD, Principal Investigator — National Hospital Organization, Mito Medical Center
Locations (1):
- Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Bunkyo-ku, Tokyo, Japan